CLINICAL TRIAL: NCT00152620
Title: Dexamethasone Versus Methylprednisolone for the Treatment of Active Inflammatory Bowel Disease
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: study completed
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 13171B
Record Dates: First submitted 2005-09-07; First posted 2005-09-09 (Estimated); Last update posted 2013-09-05 (Estimated); Status verified 2013-09

CONDITIONS: Inflammatory Bowel Disease (IBD)
Keywords: Inflammatory Bowel Disease (IBD)
MeSH Terms: conditions — Inflammatory Bowel Diseases | interventions — Dexamethasone; Methylprednisolone

INTERVENTIONS:
Drug: Dexamethasone
Drug: Methylprednisolone

SUMMARY:
The aim of this therapeutic trial is to compare the response of subjects with active IBD to daily intravenous dexamethasone versus the response to daily intravenous methylprednisolone.

ELIGIBILITY:
Inclusion Criteria:

* Parental informed consent
* Subjects 6 to 19 years of age with confirmed diagnosis of IBD (Crohn's disease, ulcerative colitis or indeterminate colitis), who on admission to the hospital have a PCDAI>15 or a Clinical-Activity Index for the Evaluation of Patients with Ulcerative Colitis of >10.
* Infectious causes (viruses, bacteria, parasites) have been ruled out.

Exclusion Criteria:

* Subjects in which the administration of corticosteroids would be contraindicated such as systemic or enteric infections diagnosed by stool analysis including culture, Clostridium Difficile toxin assay, rotavirus or adenovirus 40/41 antigens.
* Subjects with enterostomy or colostomy
* Subjects with one or more of the following conditions: unstable vital signs, acute abdomen, toxic megacolon, intestinal obstruction, intestinal perforation

Ages: 6 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40
Dates: Start 2004-06; Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
Pediatric Crohn's Disease Activity Index (PCDAI)
Clinical-Activity Index for the Evaluation of Patients with Ulcerative Colitis

SECONDARY OUTCOMES:
Partial Harvey Bradshaw score (pHB)

CONTACTS AND LOCATIONS:
Overall Officials: Barbara S Kirschner, MD, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago Comer Children's Hospital, Chicago, Illinois, United States

REFERENCES:
- [Background] EDWARDS FC, TRUELOVE SC. THE COURSE AND PROGNOSIS OF ULCERATIVE COLITIS. III. COMPLICATIONS. Gut. 1964 Feb;5(1):1-22. doi: 10.1136/gut.5.1.1. No abstract available. PMID 14127503
- [Background] Truelove SC. The management of ulcerative colitis. Br J Clin Pract. 1974 Jan;28(1):5-10. No abstract available. PMID 4149894
- [Background] Boumpas DT, Paliogianni F, Anastassiou ED, Balow JE. Glucocorticosteroid action on the immune system: molecular and cellular aspects. Clin Exp Rheumatol. 1991 Jul-Aug;9(4):413-23. PMID 1934694
- [Background] Barnes PJ, Adcock I. Anti-inflammatory actions of steroids: molecular mechanisms. Trends Pharmacol Sci. 1993 Dec;14(12):436-41. doi: 10.1016/0165-6147(93)90184-l. PMID 7510080
- [Background] Chun A, Chadi RM, Korelitz BI, Colonna T, Felder JB, Jackson MH, Morgenstern EH, Rubin SD, Sacknoff AG, Gleim GM. Intravenous corticotrophin vs. hydrocortisone in the treatment of hospitalized patients with Crohn's disease: a randomized double-blind study and follow-up. Inflamm Bowel Dis. 1998 Aug;4(3):177-81. doi: 10.1097/00054725-199808000-00001. PMID 9741018
- [Background] Truelove SC, Jewell DP. Intensive intravenous regimen for severe attacks of ulcerative colitis. Lancet. 1974 Jun 1;1(7866):1067-70. doi: 10.1016/s0140-6736(74)90552-2. No abstract available. PMID 4135487
- [Background] Stein RB, Hanauer SB. Medical therapy for inflammatory bowel disease. Gastroenterol Clin North Am. 1999 Jun;28(2):297-321. doi: 10.1016/s0889-8553(05)70058-3. PMID 10372270
- [Background] Meyers S, Lerer PK, Feuer EJ, Johnson JW, Janowitz HD. Predicting the outcome of corticoid therapy for acute ulcerative colitis. Results of a prospective, randomized, double-blind clinical trial. J Clin Gastroenterol. 1987 Feb;9(1):50-4. doi: 10.1097/00004836-198702000-00013. PMID 3031150
- [Background] Kaplan HP, Portnoy B, Binder HJ, Amatruda T, Spiro H. A controlled evaluation of intravenous adrenocorticotropic hormone and hydrocortisone in the treatment of acute colitis. Gastroenterology. 1975 Jul;69(1):91-5. PMID 168121
- [Background] Panes J, Esteve M, Cabre E, Hinojosa J, Andreu M, Sans M, Fernandez-Banares F, Feu F, Gassull MA, Pique JM. Comparison of heparin and steroids in the treatment of moderate and severe ulcerative colitis. Gastroenterology. 2000 Oct;119(4):903-8. doi: 10.1053/gast.2000.18159. PMID 11040177
- [Background] Sood A, Midha V, Sood N, Awasthi G. A prospective, open-label trial assessing dexamethasone pulse therapy in moderate to severe ulcerative colitis. J Clin Gastroenterol. 2002 Oct;35(4):328-31. doi: 10.1097/00004836-200210000-00009. PMID 12352296
- [Background] Mager DE, Lin SX, Blum RA, Lates CD, Jusko WJ. Dose equivalency evaluation of major corticosteroids: pharmacokinetics and cell trafficking and cortisol dynamics. J Clin Pharmacol. 2003 Nov;43(11):1216-27. doi: 10.1177/0091270003258651. PMID 14551176
- [Background] Campieri M. New steroids and new salicylates in inflammatory bowel disease: a critical appraisal. Gut. 2002 May;50 Suppl 3(Suppl 3):III43-6. doi: 10.1136/gut.50.suppl_3.iii43. PMID 11953332